CLINICAL TRIAL: NCT03923179
Title: The Efficacy and Safety of Pyrotinib Combined With Etoposide in HER2-positive Advanced Breast Cancer
Brief Title: Phase II Clinical Study of Pyrotinib Combined With Etoposide to Treat HER2-positive Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Li Qiao, Clinical Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LQ007
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pyrotinib+Etoposide (Experimental)
  Interventions: Drug: Pyrotinib; Drug: Etoposide

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib, 400mg qd
Drug: Etoposide — Etoposide, 50mg，qd,d1-21,Q4W

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Pyrotinib Combined With Etoposide to Treat HER2-positive Advanced Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age：18~75 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
3. A life expectancy of more than 12 weeks;
4. patients have at least one measurable lesion exists according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria and progresses after the last anti-tumor treatment or during treatment;
5. Pathologically confirmed HER2-expressing patients with locally advanced or metastatic breast cancer: HER2 IHC 3+, or HER2 IHC 2+ and FISH detection gene amplification
6. Progression after treatment with trastuzumab or treatment, patients who are no longer able to receive trastuzumab or lapatinib: continuous use of trastuzumab ≥ 2 cycles during relapse/metastasis Or during the adjuvant treatment, continuous use of trastuzumab ≥ 3 months, recurrence / metastasis after treatment or treatment;
7. echocardiography indicates that LVEF ≥ 50%;
8. The laboratory tests confirmed that the bone marrow function and liver and kidney function of the patient met the following requirements before the first dose:

   1. ANC≥1.5×10^9/L；
   2. PLT≥100×10^9/L;
   3. Hb≥100 g/L
   4. serum creatinine(Scr) less than 1.5 times the upper limit of normal value or the creatinine clearance rate calculated greater than 60 mL/min;
   5. total bilirubin less than 1.5 times the upper limit of normal value
   6. aspartate aminotransferase (AST), or alanine aminotransferase (ALT) less than 2.5 times the upper limit of normal value, less than 5 times the upper limit of normal value in patients with liver metastases;
   7. urine routine test with urinary protein more than ++, or 24 hour urinary protein more than 1.0 g;
9. Females of childbearing potential must be a pregnancy test in 7 days before participating ( including serum or urine), and the results were negative, and they are willing to take effective contraceptive methods during the trial;
10. The patient volunteered to join the study and signed an informed consent form.

Exclusion Criteria:

1. Previously treated with pyrrolidine or neratinib;
2. Previously received etoposide treatment;
3. Patients with high blood pressure who are not well controlled by antihypertensive medication (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg); have uncontrolled or severe cardiovascular disease, such as within 6 months before screening Refractory angina pectoris, congestive heart failure occurred; myocardial infarction occurred within 12 months before screening; any clinically significant ventricular arrhythmia history, QT interval prolongation; history of cerebrovascular accident, symptomatic and need Medically treated coronary heart disease;
4. having significant clinical dysfunction of the digestive tract may affect the intake, transport or absorption of oral medications (eg, inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
5. Refractory, 2 degrees and above persistent diarrhea;
6. exiting unstable brain metastasis and / or meningeal metastasis;
7. Have undergone major surgery or severe traumatic injury, fracture, or healed wound within 4 weeks;
8. Allergic to pyrotinib, etoposide and/or its excipients has been confirmed;
9. Female patients during pregnancy or lactation, female patients with fertility and positive pregnancy test, or women of childbearing age who are unwilling to take effective contraceptive measures during the whole trial period;
10. The patient has a severe concomitant disease, or any other condition that the investigator believes is not suitable for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-04-19 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | 4 months
  Refers to the proportion of patients whose tumors have shrunk to a certain proportion and maintained for a certain period of time, including cases of CR and PR, RECIST 1.1 were used to assess objective tumor remission

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | 4 months
  the date from the first dose to the first occurrence of disease progression or death from any cause, whichever occurs first
disease control rate(DCR) | 4 months
  Percentage of confirmed complete remission (CR), partial remission (PR), and disease stable (SD) cases in patients with evaluable efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Qiao I Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Binghe Xu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, ChineseAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu J, He M, Jiang M, Zhou S, Zhang M, Li Y, Chen S, Cai R, Mo H, Lan B, Ma F, Xu B, Li Q. Pyrotinib combined with metronomic etoposide in heavily pretreated HER2-positive metastatic breast cancer: a single-arm, phase II study. BMC Cancer. 2024 Oct 18;24(1):1290. doi: 10.1186/s12885-024-13041-8. PMID 39425028